CLINICAL TRIAL: NCT02809352
Title: Epidemiology of High-risk HPV Infection in Women Participating in a Pilot Screening Program Entitled START-HPV (STudy of Primary Screening in the ARdennes Department by Testing for HPV Infection)
Brief Title: Epidemiology of High-risk HPV Infection in Women Participating in a Pilot Screening Program for Cervical Cancer
Acronym: Epi-START
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PJ12078
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extraction from cervical smears (DNAPap Cervical Sampler device, Qiagen) or from self-collected vaginal lavages (Delphi-screener device, DelphiBioscience) and HPV genotyping with the Multiplex HPV Genotyping kit© (Multimetrix, Progen) based on a Luminex technology.

GROUPS / COHORTS (1):
- women tested positive for hrHPV: All women participating in START-HPV pilot program for cervical cancer screening and tested positive for hrHPV with the Hybrid Capture 2 test (Qiagen).
  Interventions: Biological: Human papillomavirus genotyping

INTERVENTIONS:
Biological: Human papillomavirus genotyping

SUMMARY:
Cervical cancer is due to a persistent infection with a group of viruses known as high-risk Human Papillomaviruses (hrHPV). Viral DNA can be easily detected in a cervical sample by a procedure called 'HPV testing', which can be used as a relevant screening test. A pilot screening program called START-HPV has been set up in the Ardennes, a French administrative area localized in the North of France, with HPV testing as a primary screening test.This observational study aimed to evaluate hrHPV genotypes repartition in the population who participate in the START-HPV screening program. This study will allow a better knowledge of hrHPV infection epidemiology in a screened population.

ELIGIBILITY:
Inclusion Criteria:

* to live in the Ardennes department (France)
* affiliation to a health insurance organism
* 31 to 65 years old

Exclusion Criteria:

* current follow-up for cervical cytological abnormalities
* history of hysterectomy
* reimbursement for a Pap smear in the last 3 years

Ages: 31 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who participate in START-HPV pilot screening program and tested positive for high-risk HPV
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HPV genotyping | Day 0
  DNA extraction from cervical smears (DNAPap Cervical Sampler device, Qiagen) or from self-collected vaginal lavages (Delphi-screener device, DelphiBioscience) and HPV genotyping with the Multiplex HPV Genotyping kit© (Multimetrix, Progen) based on a Luminex technology

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France